CLINICAL TRIAL: NCT06558630
Title: A Prospective Observational Cohort Study of Airway Management in Emergency Departments in the Netherlands.
Brief Title: ED Airway Management in the Netherlands.
Acronym: DEAR
Status: Recruiting | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: DEAR
Record Dates: First submitted 2024-04-11; First posted 2024-08-19 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Endotracheal Intubation
Keywords: Emergency department; Airway management
MeSH Terms: conditions — Emergencies | interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient in need of airway management.: All patients who undergo airway management in de ED. In this study, airway management is defined as the process of planning, preparation and execution of endotracheal intubation. While the term airway management can also be used for techniques such as placing an oropharyngeal tube, patients are only included if endotracheal intubation is attempted.
  Interventions: Procedure: Endotracheal intubation

INTERVENTIONS:
Procedure: Endotracheal intubation — Over the course of several years as many as possible ED centres in the Netherlands will be included in the collection of all data involving airway management. Airway management is defined as the process of planning, preparation and execution of endotracheal intubation.

SUMMARY:
Airway management is one of the resuscitative procedures patients may undergo in the Emergency Department (ED). While this is a high risk procedure, to date there is no data available on airway management practices, success or safety in EDs in the Netherlands. The objective of this study is to describe airway management in the Netherlands.

DETAILED DESCRIPTION:
Airway management is the planning, preparation and execution of medical interventions to maintain a patients airway and thereby maintaining or supporting the patients respiration. While the term is used for a range of techniques, the technique that is most studied and relevant in the emergency department (ED) is endotracheal intubation. Endotracheal intubation is an important procedure in emergency care with a broad range of indications. Examples are altered mental status due to trauma, intoxication or stroke, respiratory failure due to respiratory diseases such as pneumonia and airway obstruction due to trauma or allergic reactions.

While endotracheal intubation can be a lifesaving intervention, it can also result in complications such as airway trauma, aspiration, hypoxia, hypotension and cardiac arrest . Peri-intubation adverse events have been reported in 12-26% of intubations. For example, Alkhouri et al reported that ED intubations were complicated by desaturation (11.9%), hypotension (7.1%), aspiration (2.7%) and cardiac arrest (1%). These complications are relatively more frequent in the ED than in the operating room, and they also seem to result in more harm. One study reported a 38-fold higher incidence of brain damage or death as result of an airway event in the ED compared to the operating room. These differences are most likely caused by multiple factors, such as anatomical and physiological difficulties of airway management due to the underlying pathology of the ED patient, training of providers and available equipment in the ED.

Valuable information about the practice of airway management in the ED can derived from one of the large national and international ED airway registries. Examples are the National Emergency Airway Registry (NEAR), the Australia and New Zealand Emergency Department Airway Registry (ANZEDAR) and the Japanese Emergency Airway management (JEAN). These registries have described indications, providers, techniques, success and adverse events of airway management in the ED. This data has also provided insights into factors that are related with success of intubation on one hand, and the occurrence of complications on the other. For example, the NEAR registry showed that the use of video laryngoscopy was associated with a higher rate of successful intubations at the first attempt than with direct laryngoscopy in trauma patients and patients with signs of a difficult anatomical airway. In these patients the rate of oesophageal intubation was lower when video laryngoscopy was used. The ANZEDAR registry showed that intubations were more often complicated by hypotension when propofol was given as induction agent and that intubations were less often complicated by hypoxia when apnoeic oxygenation was used. Furthermore, data from these registries also show trends in the practice of airway management. For example, where only the minority of patients in the JEAN registry was intubated using rapid sequence induction (RSI) at the start of the registry, now the majority of patients is intubated using RSI. Video laryngoscopy was increasingly used during the study period in the NEAR and JEAN registries, while in the ANZEDAR registry the use of ketamine as an induction agent has significantly increased throughout the years. All in all, ED registries have provided a valuable contribution to our knowledge of ED airway management.

To date, no data has been published about airway management in EDs in the Netherlands. While the aforementioned ED registries do provide information, it is unknown to what extend those findings can be translated to the Netherlands. First of all, there is variation in the practice of airway management between the registries. For example, when comparing induction agents that are used for intubation, there is great variability between ED airway registries. In the NEAR registry etomidate was used in the great majority of intubations, while in the JEAN registry midazolam was used most often. For intubations in the ANZEDAR registry ketamine, propofol and thiopentone were used in approximately equal proportions. Considering the variations between these registries, it is difficult to make assumptions about which drugs are used in the Netherlands for airway management. Furthermore, certain features of ED care in the Netherlands differ from the countries that participated in the registries. In the NEAR, ANZEDAR and JEAN registries the intubations were mainly performed by emergency physicians. However, according to a national survey only a minority of emergency physicians in the Netherlands perform intubations. It is unclear to what extent findings of these ED registries match the current practices of airway management in EDs in the Netherlands.

The goal of this study is to provide a compressive overview of airway management practice in Dutch EDs and to provide input for quality assessment, quality improvement and future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo airway management in the ED.

Exclusion Criteria:

* ED patients that undergo airway management outside of the ED (e.g. operation room), will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patiënts who require endotracheal intubation will be included. Population will therefore be limited to those needing airway management.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events during or after endotracheal intubation | Within 10 minutes after start of procedure. The data has to reported within 24 hours of endotracheal intubation.
  The occurrence of adverse events peri-intubation, the following adverse events are defined:
  * Desaturation, defined as a decrease of SpO2 of 10% or more
  * Hypotension, defined as a systolic blood pressure of <90mmHg AND a decrease of 20% or more. In case of suspected raised intracranial pressure hypotension is defined as a systolic blood pressure of <120mmHg AND a decrease of 20% or more.
  * Hypertension
  * Bradycardia
  * Tachycardia
  * Cardiac arrest
  * Aspiration
  * Oesophageal intubation
  * Mainstem intubation
  * Dental trauma
  * Airway bleeding due to intubation attempt
  * Other adverse event, further specified by provider

SECONDARY OUTCOMES:
First pass success | Peri-intubation. The data has to reported within 24 hours of endotracheal intubation.
  The percentage of patients that are successfully intubated during the first attempt of endotracheal intubation. An attempt is defined as an attempt to visualize the larynx and an attempt ends when the laryngoscope blade is removed from the mouth.
Indications for intubation | Peri-intubation. The data has to reported within 24 hours of endotracheal intubation.
  The underlying pathology that led to the decision to intubate, these are defined as:
  * Pulmonary
  * Cardiac
  * Neurologic
  * Cardiac arrest
  * Post-cardiac arrest
  * Intoxication
  * Metabolic derangement
  * Trauma
  * Shock
  * Airway obstruction
  * Other

CONTACTS AND LOCATIONS:
Locations (1):
- Leeuwarden Medical Centre, Leeuwarden, Netherlands